CLINICAL TRIAL: NCT01840956
Title: A Phase I Study for the Evaluation of Safety and Efficacy of Humacyte's Human Acellular Vascular Graft for Use as a Vascular Prosthesis for Hemodialysis Access in Patients With End-Stage Renal Disease
Brief Title: Safety and Efficacy of a Vascular Prosthesis for Hemodialysis Access in Patients With End-Stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Aptiv Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V003
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: End-stage Renal Disease; Kidney Failure, Chronic
Keywords: End-stage Renal Disease; Hemodialysis; Chronic Renal Insufficiency; Renal Dialysis; Hemodiafiltration; Blood Vessel Prosthesis; Tissue-Engineered Vascular Graft; Vascular Prosthesis Implantation; Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency; Urologic Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Kidney Diseases; Renal Insufficiency; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAVG (Experimental): Surgical placement of HAVG
  Interventions: Biological: HAVG

INTERVENTIONS:
Biological: HAVG — HAVG is implanted into patients' arm.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a novel, tissue-engineered vascular prosthesis, the Human Acellular Vascular Graft, HAVG.

The HAVG is intended as an alternative to synthetic materials and to autologous grafts in the creation of vascular access for dialysis.

DETAILED DESCRIPTION:
The HAVG is a sterile, non-pyrogenic, acellular tubular graft composed of human collagens and other natural extra-cellular matrix proteins. Upon implantation, it is anticipated (based on pre-clinical studies) that the collagen-based matrix comprising the graft will be infiltrated with host cells and re-modeled by the host. This will result in a vascular structure more similar to the histological composition of the native vascular tissue that may improve graft longevity and be less likely to become infected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD who are not, or who are no longer candidates for creation of an autologous AV fistula and therefore need placement of an AV graft in the upper extremity to start or maintain hemodialysis therapy
* Age 18 to 80 years old, inclusive
* Suitable anatomy for implantation of straight forearm grafts or curved upper arm grafts (arterial anastomosis to radial or brachial artery, venous anastomosis to either brachial cephalic or very central basilica vein)
* Hemoglobin ≥8 g/dL and platelet count ≥100,000 cells/mm3 prior to Day 1
* Other hematological and biochemical parameters within a range consistent with ESRD and acceptable for the administration of general anesthesia prior to Day 1
* Adequate liver function, defined as serum bilirubin ≤1.5 mg/dL; GGT, AST, ALT, and alkaline phosphatase ≤2x upper limit of normal or international normalized ratio (INR) ≤1.5 prior to Day 1.
* Able to communicate meaningfully with investigative staff, competent to give written informed consent, and able to comply with entire study procedures
* Able and willing to give informed consent
* Life expectancy of at least 1 year

Exclusion Criteria:

* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within 6 months of study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Uncontrolled or poorly controlled diabetes; hospitalization for poor glucose control within the previous 6 months is an absolute exclusion criterion
* History or evidence of severe peripheral vascular disease in the upper limbs
* Known or suspected central vein obstruction on the side of planned graft implantation
* Stroke within 6 months of study entry (Day 1)
* Candidate for renal transplantation
* Treatment with any investigational drug or device within 60 days prior to study entry (Day 1)
* Treatment with vitamin K-antagonists, factor Xa inhibitors, or direct thrombin inhibitors within the month prior to study entry (Day 1)
* Female patients who are pregnant, intending to become pregnant, nursing or intending to nurse during the study
* Female patients of child bearing potential (not surgically sterile or at least 2 years post menopause) who do not use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly), eg, implants, injectables, combined oral contraceptives in combination with a barrier method, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
* History of cancer with active disease or treatment within the previous year
* Immunodeficiency including AIDS / HIV
* Documented hypercoagulable state or history of 2 or more DVTs or other spontaneous intravascular thrombotic events (thromboses of previous dialysis accesses do not count)
* Bleeding diathesis
* Active clinically significant autoimmune disease
* History of heparin-induced thrombocytopenia
* Previous PTFE graft in the operative limb unless the HAVG can be placed more proximally than the previous failed graft
* More than 1 failed PTFE graft in the operative limb
* Active local or systemic infection (WBC > 15,000 cells/mm3)
* Patients receiving a forearm graft with which crosses the elbow
* Patients receiving an upper arm graft with arterial anastomosis to the axillary artery or venous anastomosis to the axillary vein unless low in the axilla and accessible for ultrasound monitoring and compression
* Patients receiving a lower extremity AV access
* Known serious allergy to aspirin
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the HAVG
* Previous enrollment in this study
* Employees of the sponsor or patients who are employees or relatives of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2016-04-28 (Actual); Study Completion 2016-04-28 (Actual)

PRIMARY OUTCOMES:
HAVG graft assessment | From baseline to week 26 after HAVG implantation.
  The incidence of aneurysm formation, anastomotic bleeding or rupture, graft infection and irritation/inflammation/infection at the implantation site will be assessed by Doppler ultrasound and tabulated.
HAVG patency rate | at Week 26 after HAVG implantation
  Determine the patency (primary, primary assisted and secondary) rate of the Humacyte HAVG by Doppler ultrasound.
Adverse Events | From baseline to week 26 after HAVG implantation.
  Frequency and severity of AEs of each patient will be documented.
HAVG graft interventions | From baseline to week 26 after HAVG implantation.
  Graft interventions of each patient will be documented.

SECONDARY OUTCOMES:
Change from baseline in Panel Reactive Antibody | From baseline to day 29, weeks 12 and 26 after HAVG implantation.
  Assess changes in the Panel Reactive Antibody response over the 6 months after graft implantation.
Development of IgG antibodies | From baseline to day 29, weeks 12 and 26 after HAVG implantation.
  Determine whether IgG antibodies to the extracellular matrix material are formed in response to implantation of the HAVG.
Graft interventions | At each visit, i.e. day 1, day 4-7, day 15, day 29, day 57, week 12, week 16, 20, 26 after HAVG implantation.
  Determine the rates of interventions needed to maintain / restore patency in the graft.
HAVG patency rates | at 12, 18, 24 months after HAVG implantation.
  Patency rates (primary, primary assisted, and secondary)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda H Szczech, MD, MSCE, Study Director — Humacyte, Inc.
Locations (3):
- United States (3):
  - Duke University Medical Center Department of Vascular Surgery, Durham, North Carolina
  - The Methodist Hospital, Houston, Texas
  - Sentara Norfolk General Hospital Vascular & Transplant Specialists, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lawson JH, Glickman MH, Ilzecki M, Jakimowicz T, Jaroszynski A, Peden EK, Pilgrim AJ, Prichard HL, Guziewicz M, Przywara S, Szmidt J, Turek J, Witkiewicz W, Zapotoczny N, Zubilewicz T, Niklason LE. Bioengineered human acellular vessels for dialysis access in patients with end-stage renal disease: two phase 2 single-arm trials. Lancet. 2016 May 14;387(10032):2026-34. doi: 10.1016/S0140-6736(16)00557-2. PMID 27203778
- See also: Results of the clinical study have been published — https://pubmed.ncbi.nlm.nih.gov/27203778/